CLINICAL TRIAL: NCT04869527
Title: Simplifying Access to Full Early Atrial Diagnostics in Single Chamber ICD Patients Using the DX Lead and Continuous Home Monitoring in Brazil
Brief Title: Full Early Atrial Diagnostics in Single Chamber ICD Patients Using the DX Lead and Home Monitoring in Brazil.
Acronym: SAFE-DX-Home
Status: Active, not recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: TA118
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: BIOTRONIK ICDs with DX Technology — The BIOTRONIK DX system offers a single chamber ICD that enables sensing of atrial signals through floating atrial dipoles, using a single ventricular lead. This technology enables enhanced arrhythmia diagnosis based on atrial and ventricular electrograms and, in addition, early diagnosis and automatic transmission of AF and heart failure (HF) diagnostic data. The DX technology provides several features in a single chamber device that are usually only found in dual chamber devices, including atrial diagnostics and SVT discrimination - early detection of SAF, increased diagnostics accuracy, dual-chamber discrimination. Nevertheless, the benefits of a single chamber device are preserved: reduced lead complications, reduced procedure complexity, elimination of costs for atrial lead. The DX system also integrates with BIOTRONIK Home Monitoring, allowing physicians to remotely follow their patients' clinical and device statuses with daily updates.

SUMMARY:
To demonstrate the value and benefits of BIOTRONIK's exclusive DX technology in assessing the incidence of supraventricular arrhythmias, mainly atrial fibrillation (AF), in patients with an indication for single chamber ICDs.

Effects of the DX technology on related events, such as delivery of therapies and medical management, including eventual complications.

Extended benefits offered by DX devices when associated with daily remote monitoring, by means of BIOTRONIK's Home Monitoring Service Center (HMSC).

DETAILED DESCRIPTION:
To demonstrate the value and benefits of BIOTRONIK's exclusive DX technology in assessing the incidence of supraventricular arrhythmias, mainly atrial fibrillation (AF), in patients with an indication for single chamber ICDs.

Effects of the DX technology on related events, such as delivery of therapies and medical management, including eventual complications.

Extended benefits offered by DX devices when associated with daily remote monitoring, by means of BIOTRONIK's Home Monitoring Service Center (HMSC).

Primary Endpoint:

- First confirmed episode of AF or atrial flutter (AFL) or supraventricular tachycardia (SVT), detected and transmitted to the HMSC.

Other events of interest:

* Rate of successful transmissions received and stored on the HMSC platform;
* Hospital admissions related to cardiologic outcomes, at any time throughout the FU period;
* A composite outcome of any of the following device-related complications: Need for any lead repositioning or replacement, pneumothorax, new pericardial effusion, tamponade, procedure-related death or wound infection, within 60 days after the ICD insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for implanting of a single chamber ICD (primary or secondary prevention) according to current guidelines;
2. Sustained sinus rhythm as the current prevalent atrial rhythm;
3. Planned de novo implantation with a BIOTRONIK single chamber DX ICD system;
4. Patient is able to understand the nature of study and to provide written informed consent;
5. Patient is willing and able to perform all follow up visits at the study site;
6. Patient is willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring concept.

Exclusion Criteria:

1. Age < 18 years
2. Any limitation to contractual capability;
3. Female patients who are pregnant or breast feeding or planning pregnancy during the course of the study;
4. Known active malignant disease or recovered from malignant disease within 2 years prior to enrollment;
5. Life expectancy < 2 years;
6. Patient is participating in any other interventional clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring an ICD implant
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Atrial Flutter or Supraventricular Tachycardia | 12 months
  First confirmed episode of AF or atrial flutter (AFL) or supraventricular tachycardia (SVT), detected and transmitted to the HMSC.

SECONDARY OUTCOMES:
Successful transmission HMSC platform | 12 months
  Number of participants with successful transmissions received and stored on the HMSC platform
Cardiologic hospitalization | 12 months
  Number of participants with hospital admissions related to cardiologic outcomes, at any time throughout the FU period;
Device related complication | 60 days
  A composite outcome of any of the following device-related complications: Number of patients who need for any lead repositioning or replacement, pneumothorax, new pericardial effusion, tamponade, procedure-related death, or wound infection, within 60 days after the ICD insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos CK Kalil, M.D., Ph.D., Principal Investigator — Santa Casa de Misericórdia de Porto Alegre - Brugada Institute
Locations (2):
- Brazil (2):
  - Santa Casa de Misericórdia de Porto Alegre - Brugada Institute, Porto Alegre, Rio Grande do Sul
  - BIOTRONIK Coml Médica LTDA, São Paulo

IPD SHARING:
Plan to Share IPD: No